CLINICAL TRIAL: NCT06142968
Title: Incidence and Outcomes of Acute on Chronic Liver Failure (ACLF) in Cirrhotic Patients at Assiut University Hospitals
Brief Title: Acute on Chronic Liver Failure in Cirrhotic Patients at Assiut University Hospitals
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nardin Nadi Roshdy Saweres, Principle invistegator, Assiut University
Other Study IDs: ACLF
Record Dates: First submitted 2023-09-14; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: laboratory tests — Laboratory tests inform of Complete blood count , liver function tests , kidney function tests abdominal ultrasound

SUMMARY:
ACLF is a distinct syndrome that is different from chronic progressive hepatic decompensation. In most cases of ACLF, patients present initially with clinical manifestations of a decompensating event, usually renal impairment, worsening of abdominal ascites, jaundice or Hepatic encephalopathy (HE) and often precipitated by bacterial infection.

DETAILED DESCRIPTION:
Liver cirrhosis is the result of progressive fibrosis in patients with chronic liver disease of any etiology, and is associated with a poor prognosis, once hepatic decompensation starts.

Cirrhosis has two main phases: the compensated phase, where patients maintain preserved liver synthetic function and have no significant extrahepatic organ impairment; this is to be compared with a decompensated phase, where increasing ascites and loss of liver synthetic function, together with presentation with other organ impairment, are common clinical presentations. Renal failure, hepatic encephalopathy (HE), recurrent infections and upper gastrointestinal bleeding from worsening portal hypertension are considered end- stage complications of decompensated cirrhosis. The term acute- on- chronic liver failure (ACLF) is used to describe the clinical syndrome where acute hepatic decompensation leads to organ failures in the setting of liver cirrhosis.

Although there is not a universal agreement about the definition of acute on chronic liver failure (ACLF), there is a wide agreement that ACLF is a distinct syndrome that is different from chronic progressive hepatic decompensation. In most cases of ACLF, patients present initially with clinical manifestations of a decompensating event, usually renal impairment, worsening of abdominal ascites, jaundice or Hepatic encephalopathy (HE) and often precipitated by bacterial infection.

In the CANONIC study, ACLF was defined as 'an acute deterioration of pre- existing chronic liver disease, sometimes related to a clear precipitating event, and associated with increased mortality at 28 days.

The North American consortium for studying liver disease (NACSELD) proposed another definition of ACLF that defines it as 'a condition in patients with underlying chronic liver disease with or without cirrhosis that is associated with mortality within 3 months in the absence of treatment of the underlying liver disease, liver support, or liver transplantation'.

Currently, the term ACLF is still a relatively new entity that has not been very well studied or investigated in our medical research environment. There are no major studies that aimed at looking at the incidence of ACLF in our medical settings.

ELIGIBILITY:
Inclusion Criteria:

* all cirrhotic patients who will be admitted to our intensive care unit in our hospital meeting the criteria of defention of ACLF according to the CANONIC trial and The European Association for the Study of the Liver graded with chronic liver failure organ failure scor ( CLIF-OF )

Exclusion Criteria:

* 1- children less than 16 years 2- adult more than 70 years 3- patients with Hepatocellular carcinoma 4- patients known to be Chronic kidney disease

Ages: 16 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all patients with liver cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
CHILD Pugh score | baseline
  Child-Pugh A: 5 to 6 points. Child-Pugh B: 7 to 9 points. Child-Pugh C: 10 to 15 points.

SECONDARY OUTCOMES:
ACLF score ( acute on chronic liver failure score ) | baseline
  higher scores represent bad outcomes , higher mortality

REFERENCES:
- [Result] Arroyo V, Moreau R, Kamath PS, Jalan R, Gines P, Nevens F, Fernandez J, To U, Garcia-Tsao G, Schnabl B. Acute-on-chronic liver failure in cirrhosis. Nat Rev Dis Primers. 2016 Jun 9;2:16041. doi: 10.1038/nrdp.2016.41. PMID 27277335
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27277335/